CLINICAL TRIAL: NCT01671514
Title: Effects of Epicatechin-enriched Dark Chocolate on Mitochondrial Function and Exercise Capacity in Patients With Both Diabetes and Heart Failure and in Sedentary Individuals
Brief Title: Effects of Dark Chocolate on Exercise Capacity, and Mitochondrial Structure and Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: The Hershey Company (Industry)
Responsible Party: Principal Investigator, Pam Taub, MD, Assistant Professor of Medicine, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: UCSD IRB 111680
Record Dates: First submitted 2012-08-20; First posted 2012-08-23 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Heart Failure; Type 2 Diabetes
Keywords: mitochondrial biogenesis; skeletal muscle; epicatechin
MeSH Terms: conditions — Heart Failure; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sedentary (Experimental): The sedentary arm will be randomly assigned to either epicatechin-enriched dark chocolate or low-epicatechin dark chocolate as a placebo. Participants will take one square of chocolate per day for 90 days.
  Interventions: Dietary Supplement: Epicatechin-enriched dark chocolate; Other: Low-epicatechin dark chocolate
- Heart failure/diabetes (Experimental): The heart failure/diabetes arm will be randomly assigned to either epicatechin-enriched dark chocolate or low-epicatechin dark chocolate as a placebo. Participants will take one square of chocolate per day for 90 days.
  Interventions: Dietary Supplement: Epicatechin-enriched dark chocolate; Other: Low-epicatechin dark chocolate

INTERVENTIONS:
Dietary Supplement: Epicatechin-enriched dark chocolate — For experimental purposes, subjects will take one square of epicatechin-enriched dark chocolate per day for 90 days.
Other: Low-epicatechin dark chocolate — As a placebo control, subjects will take 1 square of low-epicatechin chocolate per day for 90 days.

SUMMARY:
The major goal of this study is to characterize the ability of dark chocolate enriched in epicatechin (a component of dark chocolate) to improve the structural and functional features of mitochondria in two groups

1. Patients with heart failure (HF) and type 2 diabetes (DM2) and
2. Normal yet sedentary individuals with impaired baseline exercise capacity (as assessed by VO2 max)

We propose that a 3 month treatment with dark chocolate will lead to a significant improvement in exercise capacity which will be secondary to the improvement in skeletal muscle structure from epicatechin.

DETAILED DESCRIPTION:
The flavanol epicatechin (which is derived from cocoa and has no known toxicity in humans) has been shown in clinical trials to increase levels of nitric oxide (NO) as assessed by flow-mediated dilation (FMD) in the brachial artery and measurements of circulating NO in plasma. NO is thought to be an activator of PGC-1 alpha [PPAR (peroxisome proliferator-activated receptor) alpha coactivator 1] which stimulates mitochondrial biogenesis. In both patients with heart failure and diabetes there is nitric oxide deficiency and mitochondrial dysfunction. In our proposed double-blinded placebo controlled clinical trial, we will test the hypothesis that chronic administration of epicatechin to patients with both heart failure and diabetes will increase levels of NO and PGC-1 alpha leading to increased mitochondrial biogenesis and improved mitochondrial function. We believe similar changes will occur in sedentary individuals.

In a preliminary study with 5 patients with heart failure and diabetes (conducted under UCSD IRB protocol number #090688) we have shown that epicatechin enriched dark chocolate improves mitochondrial structure (Taub PR, Ramirez-Sanchez I, Ciaraldi TP, et al. Alterations in Skeletal Muscle Indicators of Mitochondrial Structure and Biogenesis in Patients with Type 2 Diabetes and Heart Failure: Effects of Epicatechin Rich Cocoa. Clin Transl Sci. 2011;5(1):43-47.)

ELIGIBILITY:
Healthy, sedentary individuals:

Inclusion Criteria:

* Healthy, inactive individuals
* BMI 27-32

Exclusion Criteria:

* Smoking or quit smoking less than 1 year prior to enrollment
* Currently taking Coumadin or Pradaxa.

Heart failure and diabetes patients:

Inclusion Criteria:

* Medically diagnosed with heart failure and diabetes
* No significant HbA1C fluctuations in past 6 months

Exclusion Criteria:

* Currently taking Insulin
* Currently taking Coumadin or Pradaxa.
* Smoking or quit smoking less than 1 year prior to enrollment

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2012-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in exercise capacity | Baseline and 3 months
  Objectively evaluate exercise capacity through cycle ergometry to measure VO2 max.
Change from baseline in skeletal muscle metabolism | Baseline and 3 months
  The change in skeletal muscle metabolism will be evaluated by magnetic resonance spectroscopy
Change from baseline in pre-specified biomarker levels in blood, skeletal muscle, and urine | Baseline and 3 months
  Skeletal muscle biopsies and blood draws will be performed to obtain experimental samples.

OTHER OUTCOMES:
Change from baseline in quality of life, health, and nutrition questionnaires | Baseline and 3 months
  Specific questionnaires utilized include SF-36 questionnaire, Morisky Medication Adherence Scale (MMAS-8) questionnaire, the Minnesota Living with Heart Failure scale (MLHFQ), the Physical Activity Enjoyment Scale (PACES), the Leisure Time Exercise questionnaire (LTE), the Multidimensional Fatigue Symptom Inventory (MFSI) and the Block Questionnaires for Dietary Fat Screening and Fruit/Vegetable/Fiber Screening

CONTACTS AND LOCATIONS:
Overall Officials: Pam Taub, MD, Principal Investigator — Assistant Professor of Medicine, University of California, San Diego
Locations (1):
- University of California, San Diego, La Jolla, California, United States

REFERENCES:
- [Background] Taub PR, Ramirez-Sanchez I, Ciaraldi TP, Perkins G, Murphy AN, Naviaux R, Hogan M, Maisel AS, Henry RR, Ceballos G, Villarreal F. Alterations in skeletal muscle indicators of mitochondrial structure and biogenesis in patients with type 2 diabetes and heart failure: effects of epicatechin rich cocoa. Clin Transl Sci. 2012 Feb;5(1):43-7. doi: 10.1111/j.1752-8062.2011.00357.x. Epub 2011 Nov 7. PMID 22376256